CLINICAL TRIAL: NCT02999152
Title: Validation of Radio-induced Damage Biomarkers : BIOM-DRI Study
Brief Title: Validation of Radio-induced Damage Biomarkers
Acronym: BIOM-DRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low rythm of inclusions, financial support terminated
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Recherche Biomedicale des Armees (Other Government); Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0901; 2016-A01446-45 (Other: ANSM)
Record Dates: First submitted 2016-09-21; First posted 2016-12-21 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Bone Metastasis; Malignant Hemopathy
Keywords: Bio-markers; Radiation; Appropriate therapeutic strategy; Total Body Irradiation; Partial Body Irradiation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Body Irradiation (Experimental): Patient suffering from a malignant blood disease that requires a total body radiation, without (or prior to) a concomitant chemotherapy, according to the following protocol: 2x2 Gray per day, for 3 days. Blood and urines samples will be performed at days 0, 1, 2 and 3 of the treatment plan.
  Interventions: Other: blood and urines samples
- Partial Body Irradiation (Experimental): Patient with at least one bone metastasis localized at the pelvis and requiring partial body radiation therapy without associated chemotherapy, according to the following protocol: 4 Gray per day for 5 days will perform blood and urines samples at days 0, 1, 2 and 3 after the beginning of the radiation treatment.
  Interventions: Other: blood and urines samples

INTERVENTIONS:
Other: blood and urines samples — For all patients the blood samples must be organized: Before, 4 hours (+/-30 min), 1 day, 2 days, and 3 days after the start of the radiation therapy.
  Collections of urine must be organized: Before, 1 day, and 2 days after the radiation therapy.

SUMMARY:
The aim of this study is to confirm in humans the relevance and the kinetics of radio-induced bio-markers in plasma and urines, previously described at the preclinical stage.

DETAILED DESCRIPTION:
The nuclear and radiologic risks monitoring is a major preoccupation for our society. During an accident, it is primordial to define the biologic dosimetry. The dose and distribution knowledge is crucial for the medical care. Indeed, Total Body Irradiation (TBI) and Partial Body Irradiation (PBI) do not have the same clinical outcome. A Total Body Irradiation induces an acute radiation syndrome with a Medullary Aplasia. A quick diagnostic would allow the optimization of the medical care.

Nowadays, the analyse of the chromosome with two centromeres is the current norm to estimate the radiation dose, but this technique is time consuming, and not adapted to an emergency situation, and to a large population.

The new genetic techniques could permit the quick radiation dosimetry diagnosis. The research of early exposition bio-markers seems to be of a major interest. These bio-markers would allow to rapidly define the radiations perceived by an exposed subject, before the apparition of the symptoms, and by the way, to conduct to a therapeutic strategy more adapted to the patient.

In this purpose, the present study will need blood and urines samples of patients totally or partially exposed to radiations, according to their usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* For the group A:

Patient suffering from a malignant blood disease requiring a whole-body radiation, without (or prior to) a concomitant chemotherapy, according to the following protocol: 2x2 Gray per day, during 3 days.

* OR For the group B:

Patient with one (or more) pelvis metastasis requiring radiation therapy without concomitant chemotherapy, according to the following protocol: 4 Gray per day for 5 days.

Exclusion Criteria:

* More than 70 years old,
* Subject presenting abnormal blood count (grade 3),
* Person with a not controlled chronic illness,
* Subject presenting an abnormal hepatic assessment (grade 3),
* Subject having already received ionizing treatments,
* Subject reached HIV, hepatitis C or any other progressive infectious diseases,
* Pregnant women or nursing mothers,
* Person under protection of justice or unable to give consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Level of haematological and biochemical markers | Day 3
  The following bio-markers levels will be calculated :
  * Blood count,
  * Pads,
  * Haemoglobin,
  * Serum iron,
  * Plasma urea,
  * Urinary urea
  * Total protein,
  * albumin
  * creatin kinase,
  * Aspartate Amino Transferase,
  * alkaline phosphatase,
  * Total cholesterol,
  * Triglycerides,
  * Plasma creatinine
  * Creatinine clearance,
  * Urinary creatinine
  * Blood glucose,
  * Citrulline,
  * erythropoietin,
  * Plasma amylase,
  * Myoglobin,
  * Troponin,
  * C reactive protein,
  * Rate of prothrombin,
  * Fibrinogen,
  * D-Dimer,
  * Factor-V,
  * Fms-like tyrosine kinase 3-Ligand.
Quantification of chromosomal aberrations | Day 3
  Quantification of chromosomal aberrations will be performed on the blood samples performed at days 0, 1, 2 and 3 after the beginning of the rays perform in the usual practice.
Detection of biochemical markers | Day 3
  The presence or absence of these markers will be notified:
  * Interleukin 1
  * Interleukin 6
  * Interleukin 8
  * Interleukin 18
  * Tumor Necrosis Factor alpha (TNF-alpha)
  * Brain-Derived Neurotrophic Factor (BDNF)
  * Granulocyte Colony-Stimulating Factor (G - CSF)
  * Serum amyloid A (SAA)
  * Growth Arrest and DNA Damage-inducible 45 (GADD45)
  * Intestinal-type Fatty Acid-Binding Protein (FABP-I)
  * Liver-type Fatty Acid-Binding Protein (L-FABP)
  * Heart-type Fatty Acid-Binding Protein (H-FABP)
  * Stem Cell Factor Receptor CD117
Metabolomics markers levels | Day 2
  The metabolomic levels of the following molecules will be calculated on urine samples:
  * 3 - Sulfate Hydroxytyrosol
  * 1, 6-Anhydro-beta-D-glucose
  * 1 - Methylnicotinamide
  * 2 - Hydroxyisobutyrate
  * 3 - aminoisobutyrate
  * 3 - hydroxyisovalerate
  * 3 - Hydroxymandelate
  * 3 - Indoxylsulfate
  * 4 - Hydroxyphenylacetate
  * Acetate
  * Acetone
  * Adipic acid
  * Alanine
  * Betaine
  * Carnitine
  * Choline
  * Cis-Aconitate
  * Citrate
  * Creatine
  * Creatinine
  * dimethylamine
  * Ethanolamine
  * Formats
  * Glucose
  * Glycine
  * Glycolate
  * Hippurate
  * Histidine
  * Hypoxanthine
  * Isethionic acid
  * Lactate
  * Methanol
  * Methylamine
  * N, N-Dimethylglycine
  * N - Acetylserotonin sulfate
  * N - Acetyltaurine
  * O - Acetylcarnitine
  * O - Phosphocholine
  * Pi-methylhistidine
  * Pyroglutamate
  * Succinate
  * Tartrate
  * Tau-methylhistidine
  * Taurine
  * Threonine
  * trans-Aconitate
  * Trigonelline
  * Trimethylamine N-oxide
  * Tyramine sulfate
  * Tyrosine
  * Tyrosol sulfate
  * Uracil
  * Robert acid
  * Valine
  * Xanthine

SECONDARY OUTCOMES:
Total dose of radiation | Day 3
  The total dose of radiation will be calculated for each patient and compared will the biologic results.
Radiation field | Day 3
  The radiation field will be define for each patient and compared with the biological results.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Magné, PhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (2):
- France (2):
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No